CLINICAL TRIAL: NCT04253470
Title: The Neverending Debate on Progesterone Elevation: Possible Solutions
Brief Title: Debate on Progesterone Elevation on the Day of Triggering
Acronym: PE
Status: Completed | Type: Observational
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: 2020xxxx
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-01

CONDITIONS: Progesterone; ART; Female Infertility; Embryo Transfer
MeSH Terms: conditions — Infertility, Female | interventions — Embryo Transfer

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cleavage stage embryo: embryo which is on day 2 or 3
  Interventions: Other: embryo transfer
- blastocyst embryo: embryo which is on day 5
  Interventions: Other: embryo transfer

INTERVENTIONS:
Other: embryo transfer — Step of the assisted reproduction in which embryos are placed into the uterus in order to obtain a pregnancy

SUMMARY:
The association between serum progesterone (P) levels, measured on the day of ovulation trigger, and the outcome of in vitro fertilization cycles, has been one of the major controversies in the field of ovarian stimulation endocrinology.

This is a single-center retrospective cohort study. Study duration period is from January 2012 to December 2016.

All fresh embryo transfer (ET) both at cleavage stage and blastocyst stage, performed in Humanitas Fertility Center during the study period, were included.

ELIGIBILITY:
Inclusion Criteria:

* All fresh embryo transfers both at cleavage stage (Day 2 and Day3) and blastocyst stage (Day 5)
* Thawed embryo transfer deriving from supernumerary embryos cycles, by P increase, by OHSS, by other reasons (i.e inadequate endometrium, medical complications, etc)

Exclusion Criteria:

* thawed embryo transfers deriving from PGTA.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: All fresh embryo transfers both at cleavage stage (Day 2 and Day3) and blastocyst stage (Day 5), and all thawed embryo transfer, except from the ones deriving from PGTA, performed from January 2012 to December 2016 in Humanitas Fertility Center were included.
Sampling Method: Non-Probability Sample
Enrollment: 8000 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2016-12-31 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Impact of PE on CPR and LBR | January 2012-December 2016
  To evaluate the impact of premature high serum P levels on the outcome of fresh embryo transfer cycles in terms of Clinical Pregnancy Rates (CPR) and Live Birth Rates (LBR).

SECONDARY OUTCOMES:
Blastocyst embryo transfers' outcomes in PE | January 2012-December 2016
  Furthermore, the present study retrospectively investigates whether the transfer of blastocysts on day 5 post-fertilization (D5-ET) may improve the CPR and the LBR in patients with P rise.

CONTACTS AND LOCATIONS:
Overall Officials: Raffaella De Cesare, Principal Investigator — Humanitas clinical and research hospital
Locations (1):
- Paolo Emanuele Levi Setti, Rozzano, MI, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] De Cesare R, Morenghi E, Cirillo F, Ronchetti C, Canevisio V, Persico P, Baggiani A, Sandri MT, Levi-Setti PE. The Role of hCG Triggering Progesterone Levels: A Real-World Retrospective Cohort Study of More Than 8000 IVF/ICSI Cycles. Front Endocrinol (Lausanne). 2020 Sep 23;11:547684. doi: 10.3389/fendo.2020.547684. eCollection 2020. PMID 33071968